CLINICAL TRIAL: NCT00359294
Title: A Phase I Multicenter, Open-label, Dose-escalating Clinical and Pharmacokinetic Study of PM00104 Administered Intravenously Over 1 Hour Daily for 5 Days, Every 3 Weeks, to Subjects With Advanced Malignant Solid Tumors or Lymphoma.
Brief Title: A Phase I Study of Zalypsis (PM00104) in Subjects With Advanced Malignant Solid Tumors or Lymphoma
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Low recruitment
Sponsor: PharmaMar (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PM104-A-002-05
Record Dates: First submitted 2006-08-01; First posted 2006-08-02 (Estimated); Results first posted 2021-07-28 (Actual); Last update posted 2021-07-28 (Actual); Status verified 2021-07

CONDITIONS: Solid Tumors; Lymphoma
Keywords: Tumor; Lymphoma; Zalypsis; PharmaMar; PM00104
MeSH Terms: conditions — Lymphoma; Neoplasms | interventions — PM 00104

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Zalypsis (PM00104) (Experimental)
  Interventions: Drug: PM00104

INTERVENTIONS:
Drug: PM00104 — Intravenously over 1 hour daily for 5 days, every 3 weeks.
  Other Names: Zalypsis

SUMMARY:
Phase I trial, dose escalating, prospective, open-label, non-randomized, multicenter study. The purpose is to determine the safety, tolerability, dose limiting toxicity (DLT) and recommended dose (RD) of PM00104, administered intravenously over 1 hour daily for 5 days every 3 weeks (this is considered as 1 cycle) to subjects with advanced malignant solid tumors or lymphoma.

DETAILED DESCRIPTION:
Phase I trial, dose escalating, prospective, open-label, non-randomized, multicenter study. The purpose is to determine the safety, tolerability, dose limiting toxicity (DLT) and recommended dose (RD) of PM00104, administered intravenously over 1 hour daily for 5 days every 3 weeks (this is considered as 1 cycle) to subjects with advanced malignant solid tumors or lymphoma. Secondary objectives are to determine the preliminary pharmacokinetics of PM00104, to evaluate the relationship between pharmacokinetics/pharmacodynamics and to evaluate the preliminary antitumor activity of PM00104. Dose-escalation guidelines will follow an accelerated phase I design for conventional cytotoxic agents in order to minimize the number of subjects treated at the subtoxic dose levels. The trial will be conducted in compliance with the protocol, Good clinical practice (GCP) and applicable regulatory requirements.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntary written informed consent of the subject obtained before any study-specific procedure.
2. Histologically or cytologically confirmed malignant solid tumor or lymphoma.
3. Subjects with malignancies that are not otherwise curable or for which no effective standard therapy exists.
4. Age ≥ 18 years.
5. Subject with measurable or non-measurable disease using the RECIST criteria
6. Recovery from any drug-related adverse event related to previous treatment, excluding alopecia and NCI-CTCAE grade < 2 peripheral neuropathy.
7. Laboratory values within 7 days prior to first infusion:

   * Platelet count ≥ 100 x109/L, hemoglobin ≥ 9 g/dL and absolute neutrophil count (ANC) ≥ 1.5 x109/L.
   * Alkaline phosphatase ≤ 2.5 x the upper limit of normal (ULN) (≤ 5 x ULN in case of extensive bone metastases)
   * Aspartate aminotransferase (AST): ≤ 2.5 x ULN
   * Alanine aminotransferase (ALT): ≤ 2.5 x ULN
   * Total bilirubin: ≤ 1.5 ULN, unless due to Gilbert's syndrome.
   * Creatinine: ≤ ULN, or calculated creatinine clearance: ≥ 60 mL/min (calculated from the Cockcroft-Gault formula; see Appendix III).
   * Albumin: ≥ 2.5 g/dL.
   * Partial thromboplastin within normal limits for the institution
   * International normalized ratio (INR) within normal limits for the institution (unless due to oral anticoagulation)
8. Performance status (ECOG) ≤ 1
9. Life expectancy ≥ 3 months.
10. Left ventricular ejection fraction (LVEF) within normal limits for the institution (LVEF of at least 50%).
11. Women of childbearing potential must have a negative serum pregnancy test before study entry. Both men and women must agree to use a medically acceptable method of contraception throughout the treatment period and for 3 months after discontinuation of treatment. Acceptable methods of contraception include complete abstinence, Intrauterine device, oral contraceptive, subdermal implant and double barrier (condom with a contraceptive sponge or contraceptive suppository).

Exclusion Criteria:

1. Prior therapy with PM00104
2. Pregnant or lactating women.
3. Less than 4 weeks from radiation therapy (8 weeks in case of extensive prior radiotherapy) or last dose of hormonal therapy, biological therapy or chemotherapy (6 weeks in case of nitrosourea, mitomycin C).
4. Prior high dose chemotherapy that needed bone marrow transplant support.
5. Subjects with untreated or uncontrolled brain or meningeal metastases.
6. Other relevant diseases or adverse clinical conditions:

   * Increased cardiac risk as defined by:

     * History or presence of unstable angina.
     * History or presence of myocardial infarction.
     * Congestive heart failure.
     * Symptomatic arrhythmia or any arrhythmia requiring ongoing treatment.
     * Abnormal ECG (i.e., patients with the following are excluded: QT prolongation-corrected QT interval > 480 msec-, signs of cardiac enlargement or hypertrophy, bundle branch block, partial bundle branch blocks, signs of ischemia or necrosis, Wolff-Parkinson-White patterns).
     * History or presence of valvular heart disease.
     * Uncontrolled arterial hypertension despite optimal medical therapy.
     * Previous mediastinal radiotherapy.
     * Previous treatment with doxorubicin at cumulative doses in excess of 400 mg/m2
   * History of significant neurological or psychiatric disorders.
   * Active infection.
   * Significant non-neoplastic liver disease (e.g., cirrhosis, chronic active hepatitis).
   * Significant non-neoplastic renal disease.
   * Immunocompromised subjects, including subjects known to be infected by human immunodeficiency virus (HIV).
   * Uncontrolled endocrine diseases (e.g., diabetes mellitus, hypothyroidism or hyperthyroidism, adrenal disorder) requiring relevant changes in medication within the last month or hospital admission within the last 3 months.
   * Any other major illness that, in the investigator's judgment, could substantially increase the risk associated with the subject's participation in this study.
7. Limitation of the subject's ability to comply with the treatment or to follow-up at a participating center. Subjects registered on this trial must be treated and followed at a participating center.
8. Treatment with any investigational product in the 30 days period prior to the first infusion.
9. Known hypersensitivity to any of the components of the drug product, including sucrose or potassium phosphate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2006-05; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Roger Bryan Cohen, MD, Principal Investigator — Fox Chase Cancer Center; Eunice Lee Kwak, MD, Principal Investigator — Massachusetts General Hospital
Locations (2):
- United States (2):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Twelve patients were enrolled and 11 patients were treated between 9 May 2006 (first consent signed) and 10 September 2008 (last follow-up). The first dose of the first cycle was administered on 15 May 2006 and the last dose of the last cycle was administered on 20 June 2008
Groups:
- Dose Level I: PM0104: 0.053 mg/m2
- Dose-level II: PM00104: 0.106 mg/m2
- Dose-level III: PM00104: 0.212 mg/m2
- Dose Level IV: PM00104: 0.318 mg/m2
- Dose Level V: PM0104: 0.475 mg/m2
Period: Overall Study
Arm/Group | Dose Level I | Dose-level II | Dose-level III | Dose Level IV | Dose Level V
Started | 1 | 1 | 3 | 4 | 3
Completed | 0 | 0 | 0 | 0 | 0
Not Completed | 1 | 1 | 3 | 4 | 3
Not completed — Progressive disease | 1 | 1 | 2 | 3 | 2
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 1
Not completed — Not treated | 0 | 0 | 0 | 1 | 0
Not completed — Physician Decision | 0 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: One patient never treated
Groups:
- Dose-level I: PM00104: 0.053 mg/m2
- Dose-level IV: PM00104: 0.318 mg/m2
- Dose-level V: PM00104: 0.475 mg/m2
- Total: Total of all reporting groups
Arm/Group | Dose-level I | Dose-level II | Dose-level III | Dose-level IV | Dose-level V | Total
Number analyzed (Participants) | 1 | 1 | 3 | 3 | 3 | 11
Age, Continuous [Median (Full Range); unit: years] | 46 [46 to 46] | 56 [56 to 56] | 54 [44 to 54] | 66.0 [58 to 68] | 57 [43 to 72] | 56 [43 to 72]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 1 | 3 | 2 | 7
  Male | 0 | 1 | 2 | 0 | 1 | 4
Race/Ethnicity, Customized [Number; unit: Participants]
  Caucasian | 1 | 1 | 3 | 3 | 2 | 10
  Asian | 0 | 0 | 0 | 0 | 1 | 1
ECOG PS [Number; unit: participants] — Eastern Cooperative Oncology Group (ECOG) performance status (PS). 0 Fully active, able to carry on all pre-disease performance without restriction; 1 Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature; 2 Ambulatory and capable of all selfcare but unable to carry out any work activities; up and about more than 50% of waking hours; 3 Capable of only limited selfcare; confined to bed or chair more than 50% of waking hours; 4 Completely disabled; cannot carry on any selfcare; totally confined to bed or chair; 5 Dead
  participants
    PS 0 | 0 | 0 | 0 | 1 | 2 | 3
    PS 1 | 1 | 1 | 3 | 2 | 1 | 8
Primary tumor [Count of Participants; unit: Participants]
  Soft tissue sarcoma | 0 | 1 | 0 | 1 | 2 | 4
  Cervix adenocarcinoma | 0 | 0 | 1 | 1 | 0 | 2
  Colorectal adenocarcinoma | 1 | 0 | 0 | 1 | 0 | 2
  Head and neck carcinoma | 0 | 0 | 1 | 0 | 0 | 1
  Pseudomyxoma peritoneii | 0 | 0 | 1 | 0 | 0 | 1
  Unknown origin | 0 | 0 | 0 | 0 | 1 | 1
Prior chemotherapy [Count of Participants; unit: Participants]
  2-5 lines | 1 | 1 | 1 | 2 | 2 | 7
  ≥ 6 lines | 0 | 0 | 2 | 1 | 1 | 4
Prior Surgery [Count of Participants; unit: Participants] | 1 | 0 | 3 | 3 | 3 | 10
Prior radiotherapy [Count of Participants; unit: Participants] | 1 | 0 | 2 | 2 | 1 | 6

OUTCOME MEASURES:

1. Primary Outcome: Patients With Dose Limiting Toxicities (DLT)
Description: DLTs were defined as follows:
  * Hematological adverse events:
    * Any grade 4 neutropenia (absolute neutrophil count (ANC) < 0.5 x109/l) for longer than five days;
    * Any grade 4 neutropenia accompanied by fever (at least 38.5°C);
    * Any grade 4 neutropenia and sepsis or other severe infection;
    * Any grade 4 thrombocytopenia.
  * Any other grade 3/4 non-hematological adverse event (AE) and any increase of cardiac troponin I ≥0.1 ng/ml together with evidence of cardiac damage by electrocardiogram (ECG) or echocardiogram (ECHO), except for untreated nausea/vomiting or hypersensitivity reactions.
  * Decrease in left ventricular ejection fraction (LVEF) > 20% compared to the patient's baseline value and/or LVEF < 50% below normal limits for the institution.
  * Delay in the initiation of a subsequent dose exceeding two weeks due to drug related AEs
Time Frame: During the first cycle (21 days)
Measure: Number; unit: participants
Arm/Group | Dose-level I | Dose-level II | Dose-level III | Dose-level IV | Dose-level V
Number analyzed (Participants) | 1 | 1 | 3 | 3 | 3
participants | 0 | 0 | 0 | 0 | 0

2. Secondary Outcome: Overall Best Tumor Response
Description: Best tumor response was defined as the best response achieved during the study according to Response Evaluation Criteria in Solid Tumors (RECIST) v1.0. Complete response (CR): disappearance of all lesions; Partial response (PR): ≥10% decrease in target lesion size or ≥15% decrease in tumor density; Disease progression (PD): ≥10% increase in target lesion size and does not meet tumor density criteria of PR density; Stable disease (SD): none of the CR, PR, or PD criteria met; RECIST,
Time Frame: every six weeks while on study, up to 2 years
Population: 11 patients were evaluable for antitumor activity
Measure: Count of Participants; unit: Participants
Arm/Group | Dose-level I | Dose-level II | Dose-level III | Dose-level IV | Dose-level V
Number analyzed (Participants) | 1 | 1 | 3 | 3 | 3
Participants
  SD | 0 | 0 | 3 | 2 | 1
  PD | 1 | 1 | 0 | 1 | 2

ADVERSE EVENTS:
Time Frame: From first infusion to study termination, up to 2 years
Description: All patients treated with PM00104 were evaluable for safety
Groups:
- PM00104: All patients were to receive treatment for at least one 3-week cycle, which consisted of PM00104 administrations daily for 5 days and all study evaluations up to the next treatment cycle. Cycles were to be repeated every three weeks until disease progression, unacceptable toxicity, intercurrent serious illness, withdrawal of informed consent by the patient, Investigator's opinion, or treatment delay > 2 weeks. Patients were considered to be on study for the duration of their treatment and for the first 30 days following treatment discontinuation, defined as the day of the last PM00104 administration
Arm/Group | PM00104
All-Cause Mortality (participants affected / at risk) | 0/11
Serious Adverse Events (participants affected / at risk) | 5/11
Other Adverse Events (participants affected / at risk) | 11/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PM00104 (N=11)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Failure to thrive (Metabolism and nutrition disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Pain in limb (Musculoskeletal and connective tissue disorders) | 1 (1)
Pancreatitis NOS (Gastrointestinal disorders) | 1 (1)
Pyrexia (Febrile Nonhaemolytic transfusion reaction) (Injury, poisoning and procedural complications) | 1 (1)
Radiation pneumonitis (Injury, poisoning and procedural complications) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PM00104 (N=11)
Abdominal discomfort (Gastrointestinal disorders) | 2 (2)
Abdominal distension (Gastrointestinal disorders) | 1 (1)
Abdominal pain NOS (Gastrointestinal disorders) | 2 (2)
Anaemia NOS (Blood and lymphatic system disorders) | 3 (5)
Anorexia (Metabolism and nutrition disorders) | 7 (16)
Anxiety (Psychiatric disorders) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (5)
Breast mass NOS (Reproductive system and breast disorders) | 1 (1)
Chest pressure sensation (General disorders) | 1 (1)
Confusional state (Psychiatric disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 4 (8)
Contusion (Skin and subcutaneous tissue disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (8)
Dehydration (Metabolism and nutrition disorders) | 3 (6)
Depression (Psychiatric disorders) | 2 (3)
Diarrhoea NOS (Gastrointestinal disorders) | 4 (7)
Difficulty in micturition (Renal and urinary disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Dry eye NOS (Eye disorders) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1)
Dyspnoea NOS (Respiratory, thoracic and mediastinal disorders) | 3 (4)
Dysuria (Renal and urinary disorders) | 1 (1)
Eyelid ptosis (Eye disorders) | 1 (1)
Fatigue (General disorders) | 6 (23)
Flatulence (Gastrointestinal disorders) | 2 (2)
Groin infection (Infections and infestations) | 1 (1)
Haematoma NOS (Vascular disorders) | 1 (2)
Haematuria (Renal and urinary disorders) | 1 (1)
Headache NOS (Nervous system disorders) | 2 (2)
Herpes zoster (Infections and infestations) | 1 (1)
Hypercalcaemia (Metabolism and nutrition disorders) | 1 (3)
Hypersensitivity NOS (Immune system disorders) | 1 (2)
Hypoglycaemia NOS (Metabolism and nutrition disorders) | 1 (2)
Hypomagnesaemia (Metabolism and nutrition disorders) | 2 (11)
Hypotension NOS (Vascular disorders) | 2 (2)
Infection NOS (Infections and infestations) | 2 (3)
Influenza like illness (General disorders) | 1 (2)
Injection site pain (General disorders) | 1 (2)
Injection site reaction NOS (General disorders) | 6 (14)
Injection site vesicles (General disorders) | 1 (2)
Insomnia (Psychiatric disorders) | 2 (2)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 (2)
Lymphoedema NOS (Vascular disorders) | 1 (1)
Muscle weakness NOS (Musculoskeletal and connective tissue disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (5)
Nasopharyngitis (Infections and infestations) | 1 (2)
Nausea (Gastrointestinal disorders) | 8 (19)
Night sweats (Skin and subcutaneous tissue disorders) | 1 (2)
Palpitations (Cardiac disorders) | 1 (2)
Paraesthesia (Nervous system disorders) | 3 (6)
Pharyngitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Phlebitis NOS (Vascular disorders) | 1 (1)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Pruritus NOS (Skin and subcutaneous tissue disorders) | 1 (1)
Pyrexia (General disorders) | 4 (6)
Rash NOS (Skin and subcutaneous tissue disorders) | 2 (2)
Retching (Gastrointestinal disorders) | 1 (1)
Rhinitis NOS (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Seasonal allergy (Immune system disorders) | 1 (1)
Skin disorder NOS (Skin and subcutaneous tissue disorders) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 3 (3)
Subcutaneous nodule (Skin and subcutaneous tissue disorders) | 1 (1)
Supraventricular arrhythmia NOS (Cardiac disorders) | 1 (2)
Sweating increased (Skin and subcutaneous tissue disorders) | 2 (3)
Tachycardia NOS (Cardiac disorders) | 1 (1)
Tenderness NOS (General disorders) | 1 (2)
Thrombosis (Vascular disorders) | 1 (2)
Tongue oedema (Gastrointestinal disorders) | 1 (1)
Toothache (Gastrointestinal disorders) | 1 (1)
Tumour associated fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Tumour pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Upper respiratory tract infection NOS (Infections and infestations) | 1 (1)
Urethral obstruction (Renal and urinary disorders) | 1 (1)
Urinary frequency (Renal and urinary disorders) | 1 (3)
Urinary tract infection NOS (Infections and infestations) | 2 (2)
Urine odour abnormal (Renal and urinary disorders) | 1 (1)
Urticaria NOS (Skin and subcutaneous tissue disorders) | 1 (1)
Visual disturbance NOS (Eye disorders) | 1 (1)
Visual field defect NOS (Nervous system disorders) | 1 (1)
Vitreous detachment (Eye disorders) | 1 (2)
Vomiting NOS (Gastrointestinal disorders) | 5 (11)
Weakness (General disorders) | 1 (2)
Weight decreased (Investigations) | 3 (4)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
This phase I study was prematurely closed due to a low recruiting rate as well as to the perception that this could be an unpractical dosing schedule when compared to other schedules evaluated in the clinical development program of PM00104.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other